CLINICAL TRIAL: NCT02566889
Title: A Phase 4, Multicenter, Open-label Study of Serum Infliximab Concentrations and Efficacy and Safety of Dose Escalation in Pediatric Patients With Inflammatory Bowel Disease
Brief Title: An Efficacy and Safety Study of Infliximab Dose Escalation in Pediatric Participants With Inflammatory Bowel Disease
Acronym: ADAPT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to the inability to enroll a sufficient number of the required subject population
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108044; C0168IBD4020 (Other: Janssen Scientific Affairs, LLC); 2015-001653-32 (EudraCT Number)
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Pediatric Inflammatory Bowel Disease; Infliximab; Pediatric Participants; Pediatric Ulcerative Colitis; Pediatric Crohn's Disease; Dose Escalation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pediatric ulcerative colitis; Pediatric Crohn's disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Group (Experimental): Participants must have completed: a) recommended infliximab induction dosing regimen of 5 milligram (mg)/kilogram (kg) at Weeks 0, 2, and 6, followed by at least 1 maintenance doses of 5 mg/kg every 8 weeks (q8wk); or b) induction regimen with doses >6 mg/kg and have received at least 2 maintenance doses of 5 mg/kg q8wk with clinical response for at least 28 days after the most recent 5 mg/kg maintenance dose; or c) maintenance doses >6 mg/kg within past 6 months and at least 2 maintenance doses of 5 mg/kg q8wk with clinical response for at least 28 days after the most recent 5 mg/kg maintenance dose; d) must have lost clinical response, after first or subsequent q8wk maintenance dose of infliximab 5 mg/kg for participants who have completed the recommended infliximab induction dosing regimen or, after most recent (second or later) q8wk maintenance dose of infliximab 5 mg/kg for participants with an induction regimen with doses >6 mg/kg or with previous maintenance doses >6 mg/kg.
  Interventions: Drug: Infliximab
- Reference Group (Experimental): Participants must have completed: a) the recommended infliximab induction dosing regimen of 5 mg/kg at Weeks 0, 2, and 6, and have maintained a stable clinical response to infliximab after at least 1 maintenance doses of 5 mg/kg q8wk; or b) an induction regimen with doses >6 mg/kg and have received at least 2 maintenance doses of 5 mg/kg q8wk and have maintained clinical response for at least 28 days after the most recent 5 mg/kg maintenance dose 5 mg/kg maintenance dose; or c) maintenance doses >6 mg/kg within the past 6 months and at least 2 maintenance doses of 5 mg/kg q8wk and have maintained a clinical response for at least 28 days after the most recent 5 mg/kg maintenance dose 5 mg/kg maintenance dose.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Participants in the dose escalation group will escalate dose from infliximab 5 mg/kg q8w to 10 mg/kg q8w at the time of loss response. Participants in the reference group will be maintained on infliximab 5 mg/kg q8w.
  Other Names: Remicade

SUMMARY:
The purpose of this study is to evaluate whether trough serum infliximab concentrations at the time of loss of clinical response will identify pediatric participants with inflammatory bowel disease (IBD) who would benefit (regain clinical response) from dose escalation above the currently approved dose [5 milligram (mg)/kilogram (kg) every 8 weeks (q8wk)] and the safety of that dose escalation.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), prospective (study following participants forward in time), open-label (all people know the identity of the intervention) study of infliximab in pediatric participants with inflammatory bowel disease. The study consists of 3 Phases: screening Phase (up to 4 weeks), open-label treatment Phase (56 weeks) and follow up safety Phase (8 weeks). The duration of participation in the study for each participant is approximately up to 68 weeks (including screening period). Participants' efficacy and safety outcomes will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must have a biopsy-confirmed diagnosis of Crohn's disease (CD) or ulcerative colitis (UC) prior to study entry
* Must meet concomitant medication stability criteria as specified in protocol
* Is considered eligible according to the tuberculosis (TB) Screening criteria specified in protocol
* Must have negative stool results for enteric pathogens. Stool studies must include a stool culture and Clostridium difficile toxin assay. These must have been performed during Screening or the current episode of disease exacerbation as long as the stool studies were performed within 4 months prior to the first administration of infliximab at Week 0
* Must have screening laboratory test results as specfied in the protocol
* Must be up to date with all immunizations in agreement with current local immunization guidelines for immunosuppressed participants prior to Screening
* Must not have discontinued infliximab therapy

Exclusion Criteria:

* Must not require, or must not have required, within the 2 months prior to Screening, surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intraabdominal or pancreatic abscess requiring surgical drainage, or other conditions possibly confounding the evaluation of benefit from infliximab treatment
* Must not have presence or history of colonic or small bowel obstruction within 6 months prior to Screening, confirmed by objective radiographic or endoscopic evidence of a stricture with resulting obstruction (example, dilation of the colon or small bowel proximal to the stricture on barium radiograph or an inability to traverse the stricture at endoscopy)
* Must not have local manifestations of CD, such as fistulae, strictures, abscesses, or other disease complications for which surgery might be indicated. Enterocutaneuous fistulae for which surgery is not indicated, are allowed
* Must not have presence of a stoma
* Must not have documented short bowel syndrome (more than 100 centimeter in total of small bowel resected)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (36):
- United States (29):
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Hartford, Connecticut
  - Wilmington, Delaware
  - Atlanta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Waltham, Massachusetts
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Mineola, New York
  - New York, New York
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Fort Worth, Texas
  - Fairfax, Virginia
  - Madison, Wisconsin
- Canada (7):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Reference arm was planned only for safety analysis in participants being treated with labeled dosing of infliximab.
Groups:
- Reference Group: Participants received infliximab 5 mg/kg intravenous (IV) infusion every 8 weeks (q8wk) up to 56 weeks with a final safety visit at Week 64. Those who lost clinical response during participation in the study were eligible to cross over to the Dose Escalation Group and receive a total of 56 weeks of therapy with infliximab, which included duration of therapy while in the Reference Group prior to dose escalation.
- Dose Escalation Group: Participants received infliximab 10 mg/kg IV infusion q8wk from Week 0 to 56 with a final safety visit at Week 64.
Period: Overall Study
Arm/Group | Reference Group | Dose Escalation Group
Started | 45 | 8
Cross-over to Dose Escalation Group (This participant was counted in both arms for safety analysis.) | 1 | 0
Completed | 32 | 3
Not Completed | 13 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Other | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference Group | Dose Escalation Group | Total
Number analyzed (Participants) | 45 | 8 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.9) | 12.9 (2.7) | 13.9 (2.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 20
  Male | 29 | 4 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 37 | 7 | 44
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 4
  United States | 42 | 7 | 49

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Week 16 After Dose Escalation as Evaluated by Pediatric Crohn's Disease Activity Index (PCDAI) in Crohn's Disease (CD) Participants
Description: Clinical response was defined as Crohn's disease (CD) participants with decrease from baseline in PCDAI of greater than or equal to (>=) 15 points with total score of less than or equal to (<=) 30 points. PCDAI includes three history items (abdominal pain, number of liquid stools, general wellbeing), five physical examination items (abdominal examination, perirectal disease, extraintestinal manifestations, weight, height), and three laboratory tests (hematocrit, albumin, erythrocyte sedimentation rate). Items are scored on a three-point scale (zero, 5, or 10 points) except for hematocrit and erythrocyte sedimentation rate which are scored as zero, 2.5 or 5 points. PCDAI scores can range from zero to 125 with higher scores indicating more active disease. Data for this OM was planned to be analyzed for Dose escalation (DE) group only.
Time Frame: Week 16
Population: Analysis population included all participants who received at least one infusion of infliximab after enrollment. Here 'N' (number of participants analyzed) signifies the number of participants for whom data was available for this endpoint
Measure: Number; unit: Participants
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 5
Participants | 4

2. Primary Outcome: Clinical Response at Week 16 After Dose Escalation as Evaluated by Mayo Score in Ulcerative Colitis (UC) Participants
Description: Clinical Response as per Mayo score was defined as decrease from baseline in partial Mayo score of >= 2 points and >= 30 percent (%) and decrease in rectal bleeding sub-score by >= 1 point or achievement of an absolute sub-score of less than or equal to (<=) 1 point (for UC participants). A Partial Mayo Score which is Mayo score without endoscopy ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]) with each ranging from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Sustained Clinical Response Through 56 Weeks After Dose Escalation
Description: Sustained clinical response at Week 56 was defined as achieving clinical response per the primary OM definitions at Week 16 and maintaining clinical response at 1 year after dose escalation (Week 56). Clinical response was defined as a decrease from baseline in PCDAI of >= 15 points with total score of =< 30 points (for CD participants) and a decrease from baseline in partial Mayo score of >=2 points and >=30% and a decrease in rectal bleeding sub-score by >= 1 point or achievement of an absolute sub-score of =< point (for UC participants). Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Up to Week 56
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Change From Baseline in Abdominal Pain and Loose/Watery Stool Frequency Sub-scores of the PCDAI at Week 16 and Week 56 in CD Participants
Description: Abdominal and loose/watery stool frequency was evaluated by using the relevant sub-scores of the PCDAI. PCDAI includes three history items (abdominal pain, number of liquid stools, general wellbeing), five physical examination items (abdominal examination, perirectal disease, extraintestinal manifestations, weight, height), and three laboratory tests (hematocrit, albumin, erythrocyte sedimentation rate). Items are scored on a three-point scale (zero, 5, or 10 points) except for hematocrit and erythrocyte sedimentation rate which are scored as zero, 2.5 or 5 points. PCDAI scores can range from zero to 125 with higher scores indicating more active disease. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 and Week 56
Population: As the study was terminated early with lesser participants and lesser sample size, data for this OM was not collected.
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Abdominal Pain Using the Wong-Baker FACES Scale at Week 16 and Week 56 in CD Participants
Description: Change from baseline in abdominal pain using the Wong-Baker FACES scale at Week 16 and Week 56 in CD participants was reported. The Wong-Baker FACES Pain Scale is a pain scale that combines pictures and numbers to allow pain to be rated by children over the age of 3. The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst". The participant must choose the face that best describes how they are feeling. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 and Week 56
Population: as for outcome 1
Measure: Number; unit: Score on a scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 5
Score on a scale
  Participant 1: Change at Week 16: number analyzed (Participants) | 1
  Participant 1: Change at Week 16 | 0
  Participant 1: Change at Week 56: number analyzed (Participants) | 1
  Participant 1: Change at Week 56 | 0
  Participant 2: Change at Week 16: number analyzed (Participants) | 1
  Participant 2: Change at Week 16 | 0
  Participant 2: Change at Week 56: number analyzed (Participants) | 1
  Participant 2: Change at Week 56 | NA — Here 'NA' signified that the data at week 56 was not collected and analyzed for this participant as study was terminated early because of lesser participants and sample size.
  Participant 3: Change at Week 16: number analyzed (Participants) | 1
  Participant 3: Change at Week 16 | 0
  Participant 3: Change at Week 56: number analyzed (Participants) | 1
  Participant 3: Change at Week 56 | NA — Here 'NA' signified that the data at week 56 was not collected and analyzed for this participant as study was terminated early because of lesser participants and sample size.
  Participant 4: Change at Week 16: number analyzed (Participants) | 1
  Participant 4: Change at Week 16 | 1
  Participant 4: Change at Week 56: number analyzed (Participants) | 1
  Participant 4: Change at Week 56 | -4
  Participant 5: Change at Week 16: number analyzed (Participants) | 1
  Participant 5: Change at Week 16 | -5
  Participant 5: Change at Week 56: number analyzed (Participants) | 1
  Participant 5: Change at Week 56 | -5

6. Secondary Outcome: Change From Baseline in Absolute Stool Frequency Based on PCDAI Score at Week 16 and Week 56 in CD Participants
Description: Change from baseline in Absolute stool frequency at Week 16 and Week 56 in CD participants were reported. PCDAI includes three history items (abdominal pain, number of liquid stools, general wellbeing), five physical examination items (abdominal examination, perirectal disease, extraintestinal manifestations, weight, height), and three laboratory tests (hematocrit, albumin, erythrocyte sedimentation rate). Items are scored on a three-point scale (zero, 5, or 10 points) except for hematocrit and erythrocyte sedimentation rate which are scored as zero, 2.5 or 5 points. PCDAI scores can range from zero to 125 with higher scores indicating more active disease. An absolute stool frequency subscore of =<1 point was indicative of mild disease. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 and Week 56
Population: as for outcome 1
Measure: Number; unit: Score on a scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 5
Score on a scale
  Participant 1: Change at Week 16: number analyzed (Participants) | 1
  Participant 1: Change at Week 16 | -9
  Participant 1: Change at Week 56: number analyzed (Participants) | 1
  Participant 1: Change at Week 56 | -3
  Participant 2: Change at Week 16: number analyzed (Participants) | 1
  Participant 2: Change at Week 16 | 2
  Participant 2: Change at Week 56: number analyzed (Participants) | 1
  Participant 2: Change at Week 56 | NA — Here 'NA' signified that the data at week 56 was not collected and analyzed for this participant as study was terminated early because of lesser participants and sample size.
  Participant 3: Change at Week 16: number analyzed (Participants) | 1
  Participant 3: Change at Week 16 | -1
  Participant 3:Change at Week 56: number analyzed (Participants) | 1
  Participant 3:Change at Week 56 | NA — Here 'NA' signified that the data at week 56 was not collected and analyzed for this participant as study was terminated early because of lesser participants and sample size.
  Participant 4: Change at Week 16: number analyzed (Participants) | 1
  Participant 4: Change at Week 16 | -2
  Participant 4: Change at Week 56: number analyzed (Participants) | 1
  Participant 4: Change at Week 56 | -1
  Participant 5: Change at Week 16: number analyzed (Participants) | 1
  Participant 5: Change at Week 16 | 1
  Participant 5: Change at Week 56: number analyzed (Participants) | 1
  Participant 5: Change at Week 56 | 1

7. Secondary Outcome: Change From Baseline in Stool Frequency Sub-Score of the Partial Mayo Score at Week 16 and Week 56 in UC Participants
Description: Change from baseline in Stool frequency sub-score of the partial Mayo score at Week 16 and Week 56 in UC participants were reported. A Partial Mayo Score which is Mayo score without endoscopy ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each ranging from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). An absolute stool frequency subscore of <=1 point was indicative of mild disease. Higher scores indicate more severe disease. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 and Week 56
Population: Analysis population included all participants who received at least one infusion of infliximab after enrollment. Here 'N' (number of participants analyzed) signifies the number of participants for whom data was available for this endpoint and 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Number; unit: Score on a scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 1
Score on a scale
  Change at Week 16 | -2
  Change at Week 56: number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Rectal Bleeding Sub-Scores of the Partial Mayo Score at Week 16 and Week 56 in UC Participants
Description: Change from baseline in rectal bleeding sub-scores of the partial Mayo score at Week 16 and Week 56 in UC participants were reported. A Partial Mayo Score which is Mayo score without endoscopy ranges from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each ranging from 0 to 3 (0=normal, 1=mild, 2=moderate, 3=severe). An absolute rectal bleeding subscore of <=1 point was indicative of mild disease. Higher scores indicate more severe disease. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 and Week 56
Population: as for outcome 7
Measure: Number; unit: Score on a scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 1
Score on a scale
  Change at Week 16 | 0
  Change at Week 56: number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Abdominal Pain Using the Wong-Baker FACES Scale at Week 16 and Week 56 in UC Participants
Description: Change from baseline in Abdominal pain using the Wong-Baker FACES scale at Week 16 and Week 56 in UC participants were reported. The Wong-Baker FACES Pain Scale is a pain scale that combines pictures and numbers to allow pain to be rated by children over the age of 3. The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst". The participant must choose the face that best describes how they are feeling. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 And Week 56
Population: as for outcome 7
Measure: Number; unit: Score on scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 1
Score on scale
  Change at Week 16 | -4
  Change at Week 56: number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Absolute Stool Frequency at Week 16 and Week 56 in UC Participants
Description: Change from baseline in absolute stool frequency at Week 16 and Week 56 in UC participants were reported. Data for this OM was planned to be analyzed for the DE group only.
Time Frame: Baseline, Week 16 And Week 56
Population: as for outcome 7
Measure: Number; unit: Score on a scale
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 1
Score on a scale
  Change at Week 16 | -6
  Change at Week 56: number analyzed (Participants) | 0

11. Secondary Outcome: Correlation of Wong-Baker FACES Scale With Clinical Remission and Response at Week 16
Description: The Wong-Baker FACES Pain Scale is a pain scale that combines pictures and numbers to allow pain to be rated by children over the age of 3. The scale shows a series of faces ranging from a happy face at 0, "No hurt" to a crying face at 10 "Hurts worst". Data for this OM was planned to be analyzed for the DE group only. Statistical test of the hypothesis (regression model) was not performed due to insufficient data being collected to permit analysis.
Time Frame: Week 16
Population: As the study was terminated early with lesser participants and lesser sample size, data for this OM was not collected.
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 0

12. Secondary Outcome: Relationship Between Abdominal Pain PCDAI Sub-Score And the Wong-Baker Faces Scale For CD Participants
Description: PCDAI is validated clinical tool used to assess disease severity in pediatric CD participants. PCDAI collects information on disease-related variables:Total number of liquid stools, abdominal pain, and general well-being (scored by participants or participant's legal representative);Extra-intestinal manifestations;Physical examinations of abdominal mass, perirectal disease;Weight change, height change or, height velocity;Hematocrit;erythrocyte sedimentation rate; albumin. PCDAI score is calculated as sum of individual component scores and ranges from 0-100 points. Wong-Baker FACES Pain Scale combines pictures and numbers to allow pain to be rated by children over age of 3. Scale shows a series of faces ranging from a happy face at 0, "No hurt" to crying face at 10 "Hurts worst". Data for this OM was planned to be analyzed for the DE group only. Statistical test of the hypothesis (regression model) was not performed due to insufficient data being collected to permit analysis.
Time Frame: Week 16 and 56
Population: As the study was terminated early with lesser participants and lesser sample size, data for this OM was not collected.
Arm/Group | Dose Escalation Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Week 64
Description: The safety analysis population included all participants who received at least one infusion of infliximab after enrollment. Reference arm was planned only for safety analysis in participants being treated with labeled dosing of infliximab. One participants who had crossed-over from reference group to Dose escalation group was counted in both arms and safety is presented accordingly.
Arm/Group | Reference Group | Dose Escalation Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/9
Other Adverse Events (participants affected / at risk) | 36/45 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Group (N=45) | Dose Escalation Group (N=9)
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Group (N=45) | Dose Escalation Group (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Dry Eye (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Anorectal Disorder (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0
Faeces Soft (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Lip Swelling (Gastrointestinal disorders) | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tongue Erythema (Gastrointestinal disorders) | 1 | 0
Tooth Disorder (Gastrointestinal disorders) | 1 | 0
Tooth Impacted (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Allergy to Arthropod Bite (Immune system disorders) | 1 | 0
Food Allergy (Immune system disorders) | 1 | 0
Adenovirus Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 3 | 0
Eczema Infected (Infections and infestations) | 1 | 0
Epstein-Barr Virus Infection (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 0
Otitis Media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis Streptococcal (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0
Staphylococcal Impetigo (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Viral Infection (Infections and infestations) | 2 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 4 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 2 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb Injury (Injury, poisoning and procedural complications) | 2 | 0
Lip Injury (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
C-Reactive Protein Increased (Investigations) | 2 | 0
Faecal Calprotectin Increased (Investigations) | 1 | 0
Heart Rate Irregular (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 1
Transaminases Increased (Investigations) | 1 | 0
Vitamin D Decreased (Investigations) | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 1
Hemianopia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Asthma Exercise Induced (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne Cystic (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Warm (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Orthostatic Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated due to the inability to enroll a sufficient number of the required participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02566889/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT02566889/SAP_001.pdf